CLINICAL TRIAL: NCT03551353
Title: Checkout Procedure Before Airway Practices To Provide Clinical Practice With Video Based Feedback
Brief Title: Checkout Procedure, Airway Practices, Video Based Feedback
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, tahsin şimşek, principal investigator, Kocaeli Derince Education and Research Hospital
Other Study IDs: 2018-111
Record Dates: First submitted 2018-04-26; First posted 2018-06-11 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Anesthesia
Keywords: video feedback; checkout prosedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group before Video-assisted feedback: Ten anesthesia residents will be included in this group. Preoperative evaluation in terms of general anesthesia will be completed for a patient before anesthesia induction. After receiving informed consent from the patient resident will complete the preparations by checking the above-mentioned list (anesthesia machine, operating room desk, monitorization methods, aspirator systems, operating room gas systems, waste systems and other anesthesia equipment) then induction will be started. All these steps will be recorded with a camera system. Once the anesthetic application is completed and all stages are recorded, the video records will be evaluated in terms of ASA guideline
  Interventions: Other: Group before Video-assisted feedback
- Group after Video-assisted feedback: Before the second phase of the study, the resident will be informed about the guideline (checkout procedure) by a staff. Then induction of general anesthesia in another patient will be recorded at all stages. Once the anesthesia application is complete, the camera record will be monitored. Differences and developments or possible similar mistakes between the records will be discussed.
  Interventions: Other: Group after Video-assisted feedback

INTERVENTIONS:
Other: Group before Video-assisted feedback — Ten anesthesia residents will be included in this group. Preoperative evaluation in terms of general anesthesia will be completed for a patient before anesthesia induction. After receiving informed consent from the patient resident will complete the preparations by checking the above-mentioned list (anesthesia machine, operating room desk, monitorization methods, aspirator systems, operating room gas systems, waste systems and other anesthesia equipment) then induction will be started. All these steps will be recorded with a camera system. Once the anesthetic application is completed and all stages are recorded, the video records will be evaluated in terms of ASA guideline
  Groups: Group before Video-assisted feedback
Other: Group after Video-assisted feedback — Before the second phase of the study, the resident will be informed about the guideline (checkout procedure) by a staff. Then induction of general anesthesia in another patient will be recorded at all stages. Once the anesthesia application is complete, the camera record will be monitored. Differences and developments or possible similar mistakes between the records will be discussed.
  Groups: Group after Video-assisted feedback

SUMMARY:
Video-assisted feedback (VAF) is an educational method used by educators in various areas of medicine. It is possible to gain technical and non-technical skills for practical applications such as cardiopulmonary resuscitation and surgical procedures . VAF is an objective proof of an individual's performance because by giving feedback it provides non debatable, accurate, real-time data. By allowing awareness on certain issues it helps correcting the mistakes. Studies have shown improvement in clinical skills after VAF

DETAILED DESCRIPTION:
Video-assisted feedback (VAF) is an educational method used by educators in various areas of medicine. It is possible to gain technical and non-technical skills for practical applications such as cardiopulmonary resuscitation and surgical procedures . VAF is an objective proof of an individual's performance because by giving feedback it provides non debatable, accurate, real-time data. By allowing awareness on certain issues it helps correcting the mistakes . Studies have shown improvement in clinical skills after VAF .

Inaccurate or incomplete control of anesthesia equipment before use is associated with serious postoperative morbidity and mortality risk. For this reason, a number of control methods have been developed before the anesthesia application. This is one of these methods that checklists are created and repeated in intermittent periods.

American society of anesthesiologists (ASA) published a guideline to improve patient safety in 2008 . This guideline is summarized as mentioned below.

ASA Checklist:

1.Verify Auxiliary Oxygen Cylinder and Self-inflating Manual Ventilation Device are Available & Functioning 2: Verify patient suction is adequate to clear the airway 3: Turn on anesthesia delivery system and confirm that ac power is available 4: Verify availability of required monitors, including alarms. 5: Verify that pressure is adequate on the spare oxygen cylinder mounted on the anesthesia machine 6: Verify that the piped gas pressures are ≥ 50 psig 7: Verify that vaporizers are adequately filled and, if applicable, that the filler ports are tightly closed. 8: Verify that there are no leaks in the gas supply lines between the flowmeters and the common gas outlet 9: Test scavenging system function. 10: Calibrate, or verify calibration of, the oxygen monitor and check the low oxygen alarm.

11: Verify carbon dioxide absorbent is not exhausted 12: Breathing system pressure and leak testing. 13: Verify that gas flows properly through the breathing circuit during both inspiration and exhalation.

14: Document completion of checkout procedures. 15: Confirm ventilator settings and evaluate readiness to deliver anesthesia care. (ANESTHESIA TIME OUT)

Ten anesthesia residents will be included in this study. Preoperative evaluation in terms of general anesthesia will be completed for a patient before anesthesia induction. After receiving informed consent from the patient resident will complete the preparations by checking the above-mentioned list (anesthesia machine, operating room desk, monitorization methods, aspirator systems, operating room gas systems, waste systems and other anesthesia equipment) then induction will be started. All these steps will be recorded with a camera system. Once the anesthetic application is completed and all stages are recorded, the video records will be evaluated in terms of ASA guideline. Before the second phase of the study, the resident will be informed about the guideline by a staff. Then induction of general anesthesia in another patient will be recorded at all stages. Once the anesthesia application is complete, the camera record will be monitored. Differences and developments or possible similar mistakes between the records will be discussed. After evaluating the records -twice for each resident- the applicability and effectiveness of the VAF training course will be investigated in the direction of the results of 20 records, before and after VAF.

The aim of the study is to assess the compliance of anesthesiology and reanimation residents with the ASA guideline in Kocaeli Derince Training and Research Hospital.

ELIGIBILITY:
Inclusion Criteria:

* anesthesia residents will be included in this study

Exclusion Criteria:

* not to work in anesthesia clinic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Same ten anesthesia residents will be included in both group
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-07-05 (Estimated); Primary Completion 2018-07-15 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
Success rates of anesthesia residents after video assisted feedback (VAF) educational method | at month two after first measurement for each participant
  Researchers will record video of participants during practical application and the video will asses by the checklist that American society of anesthesiologists (ASA) published in 2008 to improve patient safety

SECONDARY OUTCOMES:
Success rates of anesthesia residents before video assisted feedback (VAF) educational method | on day 1 for each participant
  Researchers will record video of participants during practical application and the video will asses by the checklist that American society of anesthesiologists (ASA) published in 2008 to improve patient safety

CONTACTS AND LOCATIONS:
Overall Officials: tahsin md şimşek, Principal Investigator — KOCAELİ DERİNCE EĞİTİM VE ARAŞTIRMA HASTANESİ